CLINICAL TRIAL: NCT07163325
Title: A Phase 1 Multicenter, Open-Label, Dose-Escalation, Safety, Pharmacokinetic, Pharmacodynamic, and Clinical Activity Study of Orally Administered EP102 Monotherapy in Participants With Advanced Solid Tumors
Brief Title: EP102 Safety and Efficacy in METTL3 Modulation in Advanced Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Epics Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: EP102-101
Record Dates: First submitted 2025-08-05; First posted 2025-09-09 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-08

CONDITIONS: Advanced Solid Tumor (Phase 1)
Keywords: Advanced Solid Tumors; EP102

STUDY DESIGN:
Intervention Model Description: The study will follow a Bayesian optimal interval (BOIN) design.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (5):
- EP102 Dose level 1 (Experimental)
  Interventions: Drug: EP102
- EP102 Dose level 2 (Experimental)
  Interventions: Drug: EP102
- EP102 Dose level 3 (Experimental)
  Interventions: Drug: EP102
- EP102 Dose level 4 (Experimental)
  Interventions: Drug: EP102
- EP102 Dose level 5 (Experimental)
  Interventions: Drug: EP102

INTERVENTIONS:
Drug: EP102 — EP102 will be administered orally

SUMMARY:
This the first-in-human (FIH) study for the Investigational Medicinal Product (IMP) EP102, is designed to explore the maximum tolerated dose (MTD), the overall safety profile, its pharmacokinetic (PK) / pharmacodynamic (PD) profile, and an exploratory evaluation of antitumor activity in participants with advanced solid tumors, who have no available standard therapy or who have failed standard therapies.

This study will inform on recommended doses for further studies, e.g. dose optimization studies and / or efficacy and safety studies.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have a histological diagnosis of locally advanced or metastatic malignant solid tumors of one of the following cancer types:

  * ovarian cancer
  * cervical cancer
  * endometrial cancer
  * testicular cancer
  * cholangiocarcinoma
  * thyroid cancer
  * parathyroid cancer
  * adrenal cancer
  * pancreatic cancer
  * non-small-cell lung cancer (NSCLC)
  * head-and neck cancer
  * renal cell cancer
  * urethral cancer
  * bladder cancer
  * colorectal cancer
  * gastric cancer
  * esophageal cancer
  * triple-negative breast cancer
  * thymoma
  * soft tissue sarcoma
* Participants must have failed (i.e. progressed on, or been intolerant to standard treatment), or no standard treatment must exist, or they must have refused standard treatment. All participants must have received at least one prior line of systemic therapy.
* Participants must have at least one measurable lesion per RECIST v1.1.
* Participant must have a life expectancy of at least 12 weeks.

Exclusion Criteria:

* Participants with an active severe infection or unexplained fever > 38.5°C during screening or on the first day of study drug administration are excluded. However, at the Investigator's discretion, participants with tumor-related fever may be enrolled.
* Participants with known human immunodeficiency virus (HIV) infection, active hepatitis B virus (HBV) infection (hepatitis B surface antigen (HBsAg) positive in serum), or active hepatitis C virus (HCV) infection (HCV RNA positive in serum).
* Participants with known dysphagia, short-bowel syndrome, gastroparesis, or any condition that may impair the ingestion or gastrointestinal absorption of orally administered drugs.
* Pregnant or breastfeeding participants.
* Participants who have received IMP or devices in other clinical trials within four weeks before the first dose.
* Participants with prior exposure to selective METTL3 inhibitor therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2025-07-24 (Actual); Primary Completion 2027-11 (Estimated); Study Completion 2028-11 (Estimated)

PRIMARY OUTCOMES:
To assess the safety and tolerability of EP102 monotherapy | Up to 21 Days after first administration
  The incidence of adverse drug reactions (ADRs) and serious adverse drug reactions (SARs) during study period
To assess the safety and tolerability of EP102 monotherapy | Up to 21 Days after first administration
  The incidence of all treatment-emergent AEs and treatment-emergent serious adverse events (SAEs) during study period
Explore the maximum tolerated dose (MTD) and recommended doses of EP102 monotherapy for subsequent studie | Up to 21 Days after first administration
  Incidence of Dose Limiting Toxicities (DLT)

SECONDARY OUTCOMES:
To characterize the pharmacokinetic (PK) profile of EP102 | Up to 21 days after first administration
  Peak Plasma Concentration (Cmax)
To characterize the pharmacokinetic (PK) profile of EP102 | Up to 21 Days after first administration
  Area under the plasma concentration versus time curve (AUC)
To characterize the pharmacokinetic (PK) profile of EP102 | Up to 21 Days after first administration
  EP102 Halflife (t1/2)
To characterize the pharmacokinetic (PK) profile of EP102 | Up to 21 Days after first administration
  Clearance (Cl)
To characterize the pharmacokinetic (PK) profile of EP102 | Up to 21 Days after first administration
  Volume of Distribution (Vd)
To preliminarily evaluate the anti-tumor activity pharmacodynamic (PD) of EP102 monotherapy | Up to 21 days after administration and up until study end
  Efficacy evaluations for confirmed and unconfirmed tumor responses: determined according to RECIST v1.1 criteria

CONTACTS AND LOCATIONS:
Locations (8):
- Belgium (2):
  - Institut Jules Bordet, Brussels
  - Cliniques universitaires Saint-Luc, Brussels
- Czechia (2):
  - Masaryk Memorial Cancer Institute, Brno
  - Olomouc University Hospital, Olomouc
- Netherlands Cancer Institute (NKI), Amsterdam, Netherlands
- Spain (3):
  - Hospital Universitari Vall d'Hebron - Vall d'Hebron Institute of Oncology, Barcelona
  - START Madrid - CIOCC, Madrid
  - Hospital Universitario de Santiago de Compostela, Santiago de Compostela

IPD SHARING:
Plan to Share IPD: Yes
The sponsor will establish which IPD will be shared after the analysis of the study results
Supporting Information: Study Protocol
Time Frame: The sponsor will establish when the IPD will be shared after the analysis of the study results
Access Criteria: The sponsor will establish the IPD access criteria after the analysis of the study results

REFERENCES:
- [Background] Dutheuil G, Oukoloff K, Korac J, Lenoir F, El Bousmaqui M, Probst N, Lapin A, Nakhabina G, Sorlet C, Parmentier N, Karila D, Ghavtadze N, Casault P, Claridge S, Sapmaz S, Slater MJ, Fraser GL. Discovery, Optimization, and Preclinical Pharmacology of EP652, a METTL3 Inhibitor with Efficacy in Liquid and Solid Tumor Models. J Med Chem. 2025 Feb 13;68(3):2981-3003. doi: 10.1021/acs.jmedchem.4c02225. Epub 2025 Jan 30. PMID 39883878